CLINICAL TRIAL: NCT06763835
Title: Development and Validation of Diagnostic and Prognostic Model of Acute Coronary Syndrome Caused by Plaque Erosion Using Novel Serum Biomarkers
Brief Title: Novel Serum Biomarkers for Identifying Plaque Erosion in ACS and Predicting Prognosis
Acronym: NBPE-ACS
Status: Active, not recruiting | Type: Observational
Sponsor: Xuebo Liu (Other)
Responsible Party: Sponsor-Investigator, Xuebo Liu, Medical Doctor, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Other Study IDs: TJH-2023-010; ITJ(QN)2203 (Other Grant/Funding Number: Clinical Research Project of Tongji Hospital of Tongji University); 18411950300 (Other Grant/Funding Number: Shanghai Science and Technology Committee)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Plaque Rupture; Acute Coronary Syndromes
Keywords: plaque erosion; plaque rupture; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Five milliliter of the participants peripheral blood were collected and tested for DNA methylation and RNA sequencing, as well as proteomics tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- acute coronary syndrome casued by plaque erosion(PE-ACS): acute coronary syndrome patients casued by plaque erosion as identified by invasive optical coherence tomography in catheter labs.(PE-ACS)
  Interventions: Diagnostic Test: Blood is drawn to test for specific biomarkers
- acute coronary syndrome casued by plaque rupture(PR-ACS): acute coronary syndrome patients casued by plaque rupture as identified by invasive optical coherence tomography in catheter labs.(PR-ACS)
  Interventions: Diagnostic Test: Blood is drawn to test for specific biomarkers

INTERVENTIONS:
Diagnostic Test: Blood is drawn to test for specific biomarkers — After identifying characteristic biomarkers that can distinguish between PE-ACS and PR-ACS, we draw blood from ACS patients for testing to assist in determining whether the ACS subtype is PE-ACS or PR-ACS.

SUMMARY:
The goal of this observational study is to find novel serum biomarkers for the accurate diagnosis of plaque erosion (PE) from acute coronary syndrome (ACS) and help predicting the prognosis of PE. The main question it aims to answer is

• Whether novel serum biomarkers could facilitate the non-invasive diagnosis and prognosis prediction of PE ? Participants will be contacted at 1,2,5 year after the diagnosis of PE-ACS or other reasons of ACS.

ELIGIBILITY:
Inclusion Criteria:

people presenting with an acute coronary syndrome (ACS)-either non-ST-segment elevation myocardial infarction (NSTE-ACS); or ST-segment elevation myocardial infarction (STE-ACS), and subsequently underwent emergent coronary angiography followed by percutaneous coronary intervention (PCI). Culprit leisions were tested using optical coheren tomograpgy and pathological diagnosis(PE OR PR) were validated by 2 independent experienced core lab members.

Exclusion Criteria:

* patients younger than 18 years or older than 85 years
* patients in cardiogenic shock
* prior coronary artery bypass grafting,
* patients with corornary stent thrombosis
* patients with left main coronary disease
* patients with congestive heart failure
* patients with life-threatening arrhythmia
* patients with thrombocytopenia patients with significant hepatic or renal impairment
* patients with septicemia, leukopenia, active inflammatory or malignant disease
* other factors compromising high-quality optical coherence tomography (OCT) imaging (e.g., severe vessel tortuosity or calcification, persistent no-reflow, lesions in distal segments, or an indeterminate culprit lesion)
* Individuals unable to provide informed consent were also excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of individuals with suspected acute coronary syndrome seeking treatment at the Department of Cardiology, Tongji Hospital, Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Specific biomarkers can serve as diagnostic and prognostic indicators for subclassifying PE-ACS or PR-ACS. | From enrollment to the end of the follow-up at 1,2,5 year
  Specific biomarkers(Methylation sites, mRNA etc,.) can serve as diagnostic and prognostic indicators for subclassifying PE-ACS or PR-ACS.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongj University School of Medicine, 200333, Shanghai ,China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Johnson TW, Raber L, Di Mario C, Bourantas CV, Jia H, Mattesini A, Gonzalo N, de la Torre Hernandez JM, Prati F, Koskinas KC, Joner M, Radu MD, Erlinge D, Regar E, Kunadian V, Maehara A, Byrne RA, Capodanno D, Akasaka T, Wijns W, Mintz GS, Guagliumi G. Clinical use of intracoronary imaging. Part 2: acute coronary syndromes, ambiguous coronary angiography findings, and guiding interventional decision-making: an expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. EuroIntervention. 2019 Aug 29;15(5):434-451. doi: 10.4244/EIJY19M06_02. PMID 31258132
- [Background] Jia H, Dai J, Hou J, Xing L, Ma L, Liu H, Xu M, Yao Y, Hu S, Yamamoto E, Lee H, Zhang S, Yu B, Jang IK. Effective anti-thrombotic therapy without stenting: intravascular optical coherence tomography-based management in plaque erosion (the EROSION study). Eur Heart J. 2017 Mar 14;38(11):792-800. doi: 10.1093/eurheartj/ehw381. PMID 27578806
- [Background] Jia H, Abtahian F, Aguirre AD, Lee S, Chia S, Lowe H, Kato K, Yonetsu T, Vergallo R, Hu S, Tian J, Lee H, Park SJ, Jang YS, Raffel OC, Mizuno K, Uemura S, Itoh T, Kakuta T, Choi SY, Dauerman HL, Prasad A, Toma C, McNulty I, Zhang S, Yu B, Fuster V, Narula J, Virmani R, Jang IK. In vivo diagnosis of plaque erosion and calcified nodule in patients with acute coronary syndrome by intravascular optical coherence tomography. J Am Coll Cardiol. 2013 Nov 5;62(19):1748-58. doi: 10.1016/j.jacc.2013.05.071. Epub 2013 Jun 27. PMID 23810884